CLINICAL TRIAL: NCT03924674
Title: Standardization of Fluids in Inpatient Settings
Brief Title: SOFI: A Quality Improvement Project to Standardize Use of Intravenous Fluids in Hospitalized Pediatric Patients
Acronym: SOFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Collaborators: American Academy of Pediatrics (Other)
Responsible Party: Principal Investigator, Sahar Rooholamini, Assistant Professor, Seattle Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: AAP VIP Network SOFI study
Record Dates: First submitted 2019-04-06; First posted 2019-04-23 (Actual); Last update posted 2021-04-29 (Actual); Status verified 2021-04

CONDITIONS: Intravenous Fluids; Fluid and Electrolyte Imbalance; ADH Inappropriate
MeSH Terms: conditions — Inappropriate ADH Syndrome | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: All sites will participate in a stepped wedge cluster randomized trial. This design is helpful when simultaneous implementation of an intervention is not feasible or practical, and allows for each site to collect baseline data for comparison with post-intervention data. There will be 3 groups (or clusters) of approximately 30-40 sites each, with randomization to intervention occurring at 2 month intervals. Randomization will be stratified by: geographic region, size and baseline rate of IVF use. By the end of the project, all sites in all groups will have received the intervention toolkit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Stepped Wedge Group 1: Sept. 2019 Launch (Active Comparator): Interventions will include:
  1. Education (webinars) for physicians and nurses regarding AAP IVF guidelines, including evidence on safety of isotonic maintenance IVF
  2. Implementation of algorithms, ordersets and checklists to guide choice of IVF and clinical indications to start/stop IVF;
  3. Tools to promote discussion about timing and necessity of routine lab draws
  4. Education and feedback for physicians regarding costs and harms of routine lab testing
  Interventions: Other: Education, clinical decision support tools
- Stepped Wedge Group 2: Nov. 2019 Launch (Active Comparator): Interventions will include:
  1. Education (webinars) for physicians and nurses regarding AAP IVF guidelines, including evidence on safety of isotonic maintenance IVF
  2. Implementation of algorithms, ordersets and checklists to guide choice of IVF and clinical indications to start/stop IVF;
  3. Tools to promote discussion about timing and necessity of routine lab draws
  4. Education and feedback for physicians regarding costs and harms of routine lab testing
  Interventions: Other: Education, clinical decision support tools
- Stepped Wedge Group 3: Jan. 2020 Launch (Active Comparator): Interventions will include:
  1. Education (webinars) for physicians and nurses regarding AAP IVF guidelines, including evidence on safety of isotonic maintenance IVF
  2. Implementation of algorithms, ordersets and checklists to guide choice of IVF and clinical indications to start/stop IVF;
  3. Tools to promote discussion about timing and necessity of routine lab draws
  4. Education and feedback for physicians regarding costs and harms of routine lab testing
  Interventions: Other: Education, clinical decision support tools

INTERVENTIONS:
Other: Education, clinical decision support tools — Interventions will include:
  1. Education (webinars) for physicians and nurses regarding AAP IVF guidelines, including evidence on safety of isotonic maintenance IVF
  2. Implementation of algorithms, ordersets and checklists to guide choice of IVF and clinical indications to start/stop IVF;
  3. Tools to promote discussion about timing and necessity of routine lab draws
  4. Education and feedback for physicians regarding costs and harms of routine lab testing

SUMMARY:
Intravenous fluids (IVF) are used in hospitalized patients to replenish the fluid and electrolyte losses of patients who cannot take adequate hydration by mouth or through their gut. Inappropriate use of IVF may cause serious problems, including abnormalities in blood electrolytes such as sodium, which can lead to serious but rare neurologic harm; pain and discomfort from multiple IV insertions and subsequent complications (e.g., IV infiltration); and inadequate monitoring for adverse effects.

Investigators currently don't know what the most commonly used IVF in hospitalized pediatric patients are, and there are no national benchmark data for IVF use. The American Academy of Pediatrics published a Guideline on maintenance IVF in November 2018, which contains one major recommendation: to use isotonic (having a similar electrolyte concentration to blood plasma) maintenance IVF in medical and surgical patients 28 days to 18 years old without pre-existing serious illnesses.

This project aims to better describe and standardize the use of IVF in inpatient pediatric settings across the U.S. and evaluate the impact of an intervention bundle on maintenance IVF use. This project aims to improve health care value by reducing the number of routine laboratory draws.

In Quality Improvement research, there are three different types of measures - outcome measures, process measures and balancing measures.

In this project, the following will be used as a process measure:

The proportion of daily weight measurements for patients on maintenance IVF.

The following will be used as balancing measures:

1. There will be no increase in the number of floor-to-PICU transfers during hospitalization from baseline.
2. There will be no increase in the number of serum sodium lab results obtained from baseline.
3. There will be no increase in adverse events prompting a change in clinical management from baseline: hypertension or edema requiring a diuretic, hypertension requiring anti-hypertensive medication, and acute kidney injury (AKI) requiring renal replacement therapy (RRT)/dialysis.

DETAILED DESCRIPTION:
Study Design

All sites will participate in a stepped wedge cluster randomized trial, with 80-120 sites total. This design is helpful when simultaneous implementation of an intervention is not feasible or practical, and allows for each site to collect baseline data for comparison with post-intervention data. There will be 3 groups (or clusters) of approximately 30-40 sites each, with randomization to intervention occurring at 2 month intervals. Randomization will be stratified by: geographic region, size and baseline rate of IVF use.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥28 days and ≤18 years old at the time of admission
* Received maintenance IVF (rate greater than 10 ml/h) on hospital day #2 at 12:01 am

Exclusion Criteria:

* ICU (PICU, NICU, CICU, etc.) patients
* Patients who have never gone home from the hospital
* Patients with active adrenal, cardiac, hepatic, neurosurgical, chronic renal, heme/onc, biochemical genetic/metabolic illnesses* (*As evidenced by: (1) listing of a condition in these categories in past medical history; and/or (2) active medication related to one of these conditions)
* Patients with diabetes insipidus, DKA, severe burns
* Patients on a psychiatric hold/primary behavioral health reason for admission with no needed medical management
* Patients with voluminous watery diarrhea > 7 days

Ages: 28 Days to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 106 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Fluid Tonicity | Monthly reports will be generated each month for each participating site through study completion, approximately 9 months.
  Increase mean proportion of hours per hospital day with exclusive isotonic IVF use to ≥80% by May 2020.
Routine Labs | Monthly reports will be generated each month for each participating site through study completion, approximately 9 months.
  Decrease number of serum WBC levels (proxy for routine labs) per hospital day by 20% from baseline by May 2020.

SECONDARY OUTCOMES:
IVF duration | Monthly reports will be generated each month for each participating site through study completion, approximately 9 months.
  Decrease proportion of time (hours) on maintenance IVF during hospitalization by 10% from baseline by May 2020.

CONTACTS AND LOCATIONS:
Overall Officials: Sahar N Rooholamini, MD, MPH, Principal Investigator — Seattle Children's Hospital/Univ. of Washington
Locations (89):
- United States (89):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Community Regional Medical Center, Fresno, California
  - Loma Linda University Children's Hospital, Loma Linda, California
  - Harbor - UCLA Medical Center, Los Angeles, California
  - UCLA Mattel Children's Hospital, Los Angeles, California
  - Valley Children's Hospital, Madera, California
  - Stanford HealthCare-ValleyCare, Pleasanton, California
  - UCSF Benioff Children's Hospital, San Francisco, California
  - Valley Presbyterian Hospital, Van Nuys, California
  - John Muir Medical Center, Walnut Creek, California
  - Nemours A.I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Wolfson Children's Hosptial, Jacksonville, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Holtz Children's Hospital, Miami, Florida
  - Sacred Heart Children's Hospital, Pensacola, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Johns Hopkins All Childrens Hospital, St. Petersburg, Florida
  - Advent Health Tampa, Tampa, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Children's Hospital of Georgia, Augusta, Georgia
  - Beverly Knight Olson Children's Hospital, Navicent Health, Macon, Georgia
  - WellStar Kennestone Hospital, Marietta, Georgia
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Saint Alphonsus Medical Center, Boise, Idaho
  - St. Luke's Children's, Boise, Idaho
  - Kootenai Health, Coeur d'Alene, Idaho
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Rush University Children's Hospital, Chicago, Illinois
  - University of Illinois Hospital, Chicago, Illinois
  - Northwestern Lake Forest Hospital, Lake Forest, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Children's Hospital - Oak Lawn, Oak Lawn, Illinois
  - Advocate Children's Hospital, Park Ridge, Illinois
  - OSF Healthcare Children's Hospital of Illinois, Peoria, Illinois
  - Northwestern Central DuPage Hospital, Winfield, Illinois
  - Beacon Children's Hospital, South Bend, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Stormont Vail Health, Topeka, Kansas
  - Wesley Medical Center/Wesley Childrens Hospital, Wichita, Kansas
  - University of Kentucky, Lexington, Kentucky
  - Our Lady of the Lake Children's Hospital, Baton Rouge, Louisiana
  - The Barbara Bush Children's Hospital at Maine Medical Center, Portland, Maine
  - Anne Arundel Medical Center, Annapolis, Maryland
  - Johns Hopkins Children's Center, Baltimore, Maryland
  - St. Agnes Hospital, Baltimore, Maryland
  - Frederick Memorial Hospital, Frederick, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - C. S. Mott Children's Hospital, Ann Arbor, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Beaumont Children's Hospital, Royal Oak, Michigan
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Children's Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center Children's Hospital, Jackson, Mississippi
  - Mercy Children's Hospital-St. Louis, St Louis, Missouri
  - The Unterberg Children's Hospital, Long Branch, New Jersey
  - Shore Medical Center, Somers Point, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - University of New Mexico Children's Hospital, Albuquerque, New Mexico
  - Kravis Children's Hospital, The Mount Sinai Hospital, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - Richmond University Medical Center, Staten Island, New York
  - Maria Fareri Children's Hospital at Westchester Medical Center, Valhalla, New York
  - Akron Childrens Mahoning Valley, Youngstown, Ohio
  - Randall Children's Hospital, Portland, Oregon
  - Doernbecher Children's Hospital, Portland, Oregon
  - St. Luke's Unversity Health Network, Bethlehem, Pennsylvania
  - St. Clair Hospital, Mount Lebanon, Pennsylvania
  - Children's Hospital at Erlanger, Chattanooga, Tennessee
  - Children's Medical Center Dallas, Dallas, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - University of Texas Medical Branch- Galveston, Galveston, Texas
  - Childrens Memorial Hermann Hospital, Houston, Texas
  - Texas Children's Hospital, Houston, Texas
  - Covenant Children's Hospital, Lubbock, Texas
  - Memorial Hermann Community Hospitals, Sugar Land, Texas
  - University of Virginia Children's Hospital, Charlottesville, Virginia
  - Augusta Medical Center, Fishersville, Virginia
  - Mary Washington Hospital, Fredericksburg, Virginia
  - The Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Carilion Children's, Roanoke, Virginia
  - Mary Bridge Children's Hospital, Tacoma, Washington
  - Central Washington Hospital, Wenatchee, Washington
  - St. Mary's Hospital, Madison, Wisconsin
  - American Family Children's Hospital, Madison, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Children's Hospital of Wisconsin - Fox Valley, Neenah, Wisconsin

IPD SHARING:
Plan to Share IPD: No
All project data will be analyzed by the study team at the aggregate level and site-level data will not be made available to other researchers.

REFERENCES:
- [Background] Feld LG, Neuspiel DR, Foster BA, Leu MG, Garber MD, Austin K, Basu RK, Conway EE Jr, Fehr JJ, Hawkins C, Kaplan RL, Rowe EV, Waseem M, Moritz ML; SUBCOMMITTEE ON FLUID AND ELECTROLYTE THERAPY. Clinical Practice Guideline: Maintenance Intravenous Fluids in Children. Pediatrics. 2018 Dec;142(6):e20183083. doi: 10.1542/peds.2018-3083. PMID 30478247
- [Background] Rooholamini SN, Clifton H, Haaland W, McGrath C, Vora SB, Crowell CS, Romero H, Foti J. Outcomes of a Clinical Pathway to Standardize Use of Maintenance Intravenous Fluids. Hosp Pediatr. 2017 Dec;7(12):703-709. doi: 10.1542/hpeds.2017-0099. PMID 29162640
- [Derived] Rooholamini SN, Jennings B, Zhou C, Kaiser SV, Garber MD, Tchou MJ, Ralston SL. Effect of a Quality Improvement Bundle to Standardize the Use of Intravenous Fluids for Hospitalized Pediatric Patients: A Stepped-Wedge, Cluster Randomized Clinical Trial. JAMA Pediatr. 2022 Jan 1;176(1):26-33. doi: 10.1001/jamapediatrics.2021.4267. PMID 34779837